CLINICAL TRIAL: NCT04554628
Title: Early Prediction of Acute Kidney Injury Among Patients Admitted to Surgical ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, lecturer of anesthesia and intensive care, Tanta University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: Security forces hospital
Record Dates: First submitted 2020-09-03; First posted 2020-09-18 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury; Biomarkers
MeSH Terms: conditions — Acute Kidney Injury | interventions — Urination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary human neutrophil gelatinase-associated lipocalin (Active Comparator): Urinary human neutrophil gelatinase-associated lipocalin (U-NGAL) measurement
  Interventions: Diagnostic Test: ELISA test in urine
- Urinary human kidney injury molecule 1 (U-KIM1) (Active Comparator): Urinary human kidney injury molecule 1 (U-KIM1) measurement group
  Interventions: Diagnostic Test: ELISA test in urine

INTERVENTIONS:
Diagnostic Test: ELISA test in urine — enzyme linked immunosorbent assay technology for detection of UNGAL and UKIM1 in urine in postoperative ICU patients
  Other Names: enzyme linked immunosorbent assay technology

SUMMARY:
Early prediction of AKI can help to improve patients' outcome through early institution of the appropriate intervention, thus the current study hypothesizes that urine analysis for certain markers may provide an early knowledge about the possibility of oncoming kidney affection secondary to organ and tissue trauma affecting patients admitted to surgical ICU.

The current study tries to evaluate the value of urinary markers as early predictors of possible development of AKI in patients admitted to surgical ICU.

DETAILED DESCRIPTION:
All patients will be clinically evaluated for demographic and clinical data. Severity of injury and number of surgical interventions will be evaluated using the simplified Therapeutic Intervention Scoring System (TISS-28) and the extent of impact of associated diseases on patients' physiological and body organs' functions will be evaluated using the Acute Physiology and Chronic Health Evaluation (APACHE II) and sequential organ failure assessment (SOFA) . Higher scores indicate more severe illness and for the TISS-28 score, each therapeutic intervention will be assigned 1 to 4 points, and the points will be summed daily to obtain the overall score and higher score indicates a higher number of therapeutic interventions.

Diagnosis of AKI Development of AKI within the first 48 hours after ICU admission and its staging will be defined according to the Acute Kidney Injury Network criteria. Each stage will be defined by the extent of change in serum creatinine level (∆SCr) as follows: Mild if Scr was increased by ≥0.3 mg/ml or ∆SCr was ≥1.5-2-fold from baseline, Moderate if ∆SCr was >2-3-fold from baseline and Severe if ∆SCr was increase by >3-fold from baseline .

Laboratory investigations Blood samples will be sent for estimation of serum creatinine (SCr) . Urine samples will be sent for spot creatinine , UNGAL, KIM1.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted to surgical ICU will be eligible for evaluation for inclusion and exclusion criteria.

Exclusion Criteria:

* Patients with manifest kidney disease.
* Patients had renal surgery
* Patients maintained on renal replacement therapy
* Patients had diabetic nephropathy.
* Patients had liver disease, endocrinopathies.
* Patients morbid obesity that was defined as body mass index (BMI) >35 kg/m2 .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
The ability of estimated urinary markers for prediction of patients susceptible to develop AKI. | 180 days
  The ability of UNGAL and UKIM1 to early predict acute kidney injury before the serum creatinine rises.

SECONDARY OUTCOMES:
The number of patients who developed rise of Serum Creatinine diagnostic of AKI and the extent of AKI severity | 180days
  The incidence of postoperative renal injury incidence
The best detector of acute kidney injury | 180 days
  The results of statistical analyses for the best predictor for upcoming AKI

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abosamak, Principal Investigator — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol